CLINICAL TRIAL: NCT06285357
Title: A Pilot Study to Test the Effect of the Association of Epigallocatechin Gallate (EGCG), Folic Acid and Vitamin B12 in Preventing the Persistence of Human Papilloma Virus (HPV) Infection.
Brief Title: The Effect of the Association EGCG, Folic Acid and Vitamin B12 in Preventing the Persistence of HPV Infection.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPISTOP_22
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-03

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — epigallocatechin gallate; Folic Acid; Vitamin B 12

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- treatment (Experimental)
  Interventions: Dietary Supplement: EGCG + folic acid + B12

INTERVENTIONS:
Dietary Supplement: EGCG + folic acid + B12 — EGCG + folic acid + B12
  Arms: treatment

SUMMARY:
The purpose of the study is to test the effect of the administration of a dietary supplement consisting of epigallocatechin gallate (EGCG), vitamin B12 and folic acid in the treatment of infections with papilloma virus of the cervix.

ELIGIBILITY:
Inclusion Criteria:

* HR-HPV DNA test positivity

Exclusion Criteria:

* No HSIL

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
HPV DNA test negativity | 8 months of treatment
  Percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria di Modena, Modena, Modena, Italy